CLINICAL TRIAL: NCT03007576
Title: Phase I Clinical Trial - Treatment of Knee Osteoarthritis With Autologous Mesenchymal Stromal Cell Product (RegStem)
Brief Title: Treatment of Knee Osteoarthritis With Autologous Mesenchymal Stromal Cell Product (RegStem)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMO Biomedicine Corporation (Industry)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMOCT01
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Osteoarthritis,Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RegStem (Experimental): Autologous MSC, 5×10^7 cells, one injection
  Interventions: Biological: RegStem

INTERVENTIONS:
Biological: RegStem — RegStem, 1.5 ml, one injection
  Other Names: MSC

SUMMARY:
Osteoarthritis (OA) is a common and incurable disease for the elderly in Taiwan, so it is an important mission to develop a new treatment for OA. Recently, cellular therapy is a new and popular medical treatment around the world, one of them is "Mesenchymal Stromal Cells (MSCs)". MSCs are found in many tissues of human body and play an important role for repairing, regeneration, anti-inflammatory and chondrogenesis. So, MSC product, RegStem, for osteoarthritis treatment becomes a developing target for new generation drugs.

This study is to isolate and expand MSCs(RegStem) from infrapatellar fat pad of subject. When the number of MSCs expands to 1×10^8, cell will be cryopreserved in the liquid nitrogen tank until all release tests passed. On the distribution day, cell will be thawed and injected into joint cavity of patient (5×10^7). Subjects will be monitored after MSC product infusion of seven days, one month, six months and one year. The monitoring items include the changes of knee (by appearance, X-ray and MRI of knee) and pain improvement (by questionnaire).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand and sign the informed consent form for this study
2. Grade 2~3 osteoarthritis according to the Kellgren-Lawrence grading scale with one-month X-ray
3. Age is 50~75 years old
4. Postmenopausal women
5. VAS scores in 50 to 90 mm

Exclusion Criteria:

1. Abnormal of liver and kidney: GOT and GPT > 100 IU/L, BUN >22 mg/dl and creatinine > 1.2 mg/dl.
2. Positive serology for HIV, HTLV-1/2 and syphilis
3. Women who are pregnant or breast feeding
4. Serious pre-existing medical conditions: coagulation disorders, cardiovascular diseases (arrhythmias, myocardial infarction and surgery), renal diseases (chronic renal failure), liver diseases (cirrhosis), diabetes mellitus type I, cancer history.
5. Other joint diseases: knee deformity (knee varus greater than 10 degree or valgus greater than 20 degree), rheumatic arthritis, gouty arthritis, septic arthritis, serious meniscal tear, other autoimmune arthritis.
6. Skin inflammatory of knee
7. Knee pain caused by referred pain from spine disease or hip joint disease. Knee pain combined with pain from spine disease or hip disease.
8. Immunosuppressive state
9. Subjects who were injected with hyaluronic acid and PRP in the past 6 months
10. Body mass index (BMI) greater than 30
11. Have a history of allergic reaction of any medication
12. Participation in another clinical trial or treatment within 3 months
13. Other pathologic conditions or circumstances that difficult participation in this study according to PI's evaluations

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Safety of RegStem by incidence of adverse events and changes in physical examinations, vital signs and the results of clinical lab tests. | 48 weeks
Clinical assessment of International Knee Documentation Committee (IKDC) score | 48 weeks
  Assess symptoms of knee, sport activity and function of knee

SECONDARY OUTCOMES:
Clinical assessment of Knee injury and Osteoarthritis Outcome Score (KOOS) | 48 weeks
Clinical assessment of visual analogue scale (VAS) | 48 weeks
Clinical assessment of knee X-ray | 48 weeks
Clinical assessment of knee MRI | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan